CLINICAL TRIAL: NCT05088720
Title: Comparative Study Between Two Doses of Misoprostol in Women With Incomplete First-trimester Miscarriage After Misoprostol Treatment: A Randomized Clinical Trial
Brief Title: Misoprostol for Management of Women With an Incomplete Miscarriage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aswu/354/7/19
Record Dates: First submitted 2021-10-10; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: a double-blind placebo-controlled randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a double-blind placebo-controlled randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- misoprostol 800 µg (Experimental): received misoprostol 800 µg (Misotac 200 µg tablets, SIGMA pharmaceutical) once dose sublingually
  Interventions: Drug: misoprostol 800 µg
- misoprostol 400 µg (Active Comparator): received misoprostol 400 µg (Misotac 200 µg tablets, SIGMA pharmaceutical) once dose sublingually
  Interventions: Drug: misoprostol 400 µg

INTERVENTIONS:
Drug: misoprostol 800 µg — received misoprostol 800 µg (Misotac 200 µg tablets, SIGMA pharmaceutical) once dose sublingually
  Arms: misoprostol 800 µg
Drug: misoprostol 400 µg — received misoprostol 400 µg (Misotac 200 µg tablets, SIGMA pharmaceutical) once dose sublingually
  Other Names: Active Comparator
  Arms: misoprostol 400 µg

SUMMARY:
Miscarriage is defined as the spontaneous loss of a pregnancy before 24 weeks gestation, that is, before fetal viability. The clinical signs of miscarriage are usually vaginal bleeding associated with abdominal pain and cramping. The miscarriage is named 'complete' or 'incomplete' according to whether or not tissues are retained in the uterus. If a woman has minimal bleeding but her cervix is closed, this is known as a 'threatened miscarriage. However; if the pregnancy is still inside the uterus but the cervix is open, this is described as an 'inevitable miscarriage', which it will not usually be possible to save the fetus.

DETAILED DESCRIPTION:
the aim of the study is to evaluate 2 doses with misoprostol in Women With Incomplete First-trimester Miscarriage After Misoprostol Treatment

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed incomplete induced miscarriage, less than 12 weeks' gestation.
* No known allergy to misoprostol.
* Women who will be hemodynamically stable.
* Good access to emergency facilities

Exclusion Criteria:

* Women with signs of severe infection ( fever > 38°)
* Women with severe vaginal bleeding
* Women are known to have allergies to prostaglandins
* Severe abdominal pain requiring immediate intervention

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with incomplete missed abortion
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
The number of patients with complete miscarriage at 1 week | 7 days
  The number of patients with complete miscarriage at 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No